CLINICAL TRIAL: NCT01047332
Title: A Randomized Trial Comparing the Uncovered to the Covered Wallstent in the Palliation of Malignant Bile Duct Strictures
Brief Title: A Trial Comparing the Uncovered to the Covered Wallstent in the Palliation of Malignant Bile Duct Strictures
Acronym: Wallstent
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Boston Scientific Corporation (Industry)
Responsible Party: Principal Investigator, David L. Carr-Locke, MD, FRCP, Dr. David Carr-Locke, MD, FRCP, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: BS-816
Record Dates: First submitted 2010-01-08; First posted 2010-01-12 (Estimated); Results first posted 2017-04-11 (Actual); Last update posted 2017-04-11 (Actual); Status verified 2017-02

CONDITIONS: Inoperable Tumors of the Bile Duct

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Uncovered Wallstent (Active Comparator): Endoscopically-placed biliary self-expanding metal stent (SEMS) (uncovered type).
  Interventions: Device: Uncovered Wallstent
- Partially Covered Wallstent (Experimental): Endoscopically-placed biliary self-expanding metal stent (SEMS) (partially covered type).
  Interventions: Device: Partially Covered Wallstent

INTERVENTIONS:
Device: Partially Covered Wallstent — Partially covered wallstent
  Arms: Partially Covered Wallstent
Device: Uncovered Wallstent — Uncovered wallstent
  Arms: Uncovered Wallstent

SUMMARY:
The purpose of the study is to determine the best management of bile duct narrowing (stricture) due to inoperable tumors. The bile duct is a tube that carries bile formed in the liver to the small bowel to digest fats. Tumors around the bile duct can compress the duct causing pain, jaundice (yellow skin and eyes), itchy skin and fever.

DETAILED DESCRIPTION:
This is a prospective randomized trial conducted at 4 large teaching hospitals (Brigham and Women's Hospital, Massachusetts General Hospital, and Boston Medical Center, Boston, Massachusetts, and Mayo Clinic, Rochester, Minnesota).

Malignancy is determined by pathology. Cancer stage is determined by transabdominal imaging and/or endoscopic ultrasound (EUS). Written informed consent is obtained from each of the enrolled patients. The study is approved by the Institutional Review Boards at each of the participating centers.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years of age.
* Malignant bile duct stricture.
* Increased bilirubin.
* Duct stricture is ≥ 1 cm distal to the biliary hilum (bifurcation of the common hepatic duct into the right and left hepatic ducts).
* Not an operative candidate.

Exclusion Criteria:

* Unable to obtain consent.
* Unable to tolerate procedure.
* Suspected benign bile duct stricture.
* Candidate for potentially curative surgical intervention.
* Previous metallic biliary stent.
* Previous bile duct surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2002-10 (Actual); Primary Completion 2008-05 (Actual); Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David L Carr-Locke, MD, FRCP, Principal Investigator — Brigham and Women's Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Telford JJ, Carr-Locke DL, Baron TH, Poneros JM, Bounds BC, Kelsey PB, Schapiro RH, Huang CS, Lichtenstein DR, Jacobson BC, Saltzman JR, Thompson CC, Forcione DG, Gostout CJ, Brugge WR. A randomized trial comparing uncovered and partially covered self-expandable metal stents in the palliation of distal malignant biliary obstruction. Gastrointest Endosc. 2010 Nov;72(5):907-14. doi: 10.1016/j.gie.2010.08.021. PMID 21034891

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Uncovered Wallstent | Partially Covered Wallstent
Started | 61 | 68
Completed | 4 (Alive at final follow-up) | 4 (Alive at final follow-up)
Not Completed | 57 | 64
Not completed — SEMS Obstruction | 11 | 20
Not completed — Died Unobstructed | 38 | 41
Not completed — Lost to Follow-up | 8 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Uncovered Wallstent | Partially Covered Wallstent | Total
Number analyzed (Participants) | 61 | 68 | 129
Age, Continuous [Mean (Standard Deviation); unit: years] | 65 (13) | 66 (14) | 66 (14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 38 | 68
  Male | 31 | 30 | 61

OUTCOME MEASURES:

1. Primary Outcome: Time to Recurrent Biliary Obstruction
Description: Biliary obstruction is the narrowing (stricture) of the bile duct. This narrowing prevents bile, which is formed in the liver, from being carried to the small bowel to digest fats. Symptoms of biliary obstruction are pain, jaundice (yellow skin and eyes), itchy skin and fever. Time to biliary obstruction is defined as the time from the placement of the stent to the time of biliary obstruction as reported by the participant via monthly interview questions or call to a pager if symptoms of recurrent biliary obstruction developed. Participants not experiencing recurrent biliary obstruction were censored at the date of last follow-up or date of death.
Time Frame: Median follow-up of 125 days in the uncovered SEMS arm and 201 days in the partially covered SEMS arm
Population: All randomized participants.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Uncovered Wallstent | Partially Covered Wallstent
Number analyzed (Participants) | 61 | 68
days | 711 [283 to NA] — Unable to calculate upper confidence interval because the largest value in the Kaplan-Meier analysis of time to recurrent biliary obstruction was censored. | 357 [264 to 1302]
Statistical Analysis 1: Comparison: Uncovered Wallstent vs Partially Covered Wallstent; Test type: Other; p = 0.530, Log Rank

2. Secondary Outcome: Patient Survival
Description: Patient survival is defined as the date of the placement of the stent to the date of death. Participants lost to follow-up were analyzed in an intention-to-treat fashion and censored at the time of their last follow-up interview.
Time Frame: Median follow-up of 125 days in the uncovered SEMS arm and 201 days in the partially covered SEMS arm
Population: All randomized participants.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Uncovered Wallstent | Partially Covered Wallstent
Number analyzed (Participants) | 61 | 68
days | 239 [84 to 401] | 227 [99 to 365]
Statistical Analysis 1: Comparison: Uncovered Wallstent vs Partially Covered Wallstent; Test type: Other; p = 0.997, Log Rank

3. Secondary Outcome: Number of Participants With Serious Adverse Events (SAEs)
Description: Serious adverse events were defined as adverse events requiring an invasive procedure or hospitalization or resulting in death.
Time Frame: From time of stent placement to participant death or lost to follow-up (up to 1302 days)
Population: All randomized participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Uncovered Wallstent | Partially Covered Wallstent
Number analyzed (Participants) | 61 | 68
Participants | 27 | 42

4. Secondary Outcome: Number of Participants With Recurrent Biliary Obstruction Reported by Mechanism
Description: Mechanisms of recurrent biliary obstructions are defined as tumor ingrowth, tumor overgrowth, stent migration, sludge, food debris, stent failed to expand and unknown. Stents may be obstructed by more than one mechanism, therefore, the total does not add up to the number of stent obstructions in each group.
Time Frame: Median follow-up of 125 days in the uncovered SEMS arm and 201 days in the partially covered SEMS arm
Population: All randomized participants.
Measure: Number; unit: participants
Arm/Group | Uncovered Wallstent | Partially Covered Wallstent
Number analyzed (Participants) | 61 | 68
participants
  Tumor ingrowth | 8 | 6
  Tumor overgrowth | 0 | 3
  Stent migration | 0 | 6
  Sludge | 1 | 4
  Food debris in the stent | 1 | 1
  Stent failed to expand | 0 | 1
  Unknown | 2 | 2

ADVERSE EVENTS:
Time Frame: From time of stent placement to participant death or lost to follow-up (up to 1302 days).
Arm/Group | Uncovered Wallstent | Partially Covered Wallstent
Serious Adverse Events (participants affected / at risk) | 27/61 | 42/68
Other Adverse Events (participants affected / at risk) | 0/61 | 0/68
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Uncovered Wallstent (N=61) | Partially Covered Wallstent (N=68)
Recurrent biliary obstruction (Hepatobiliary disorders) | 15 | 34
Stent migration (General disorders) | 0 | 8
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 3 | 3
Pain (General disorders) | 6 | 6
Line infection (Infections and infestations) | 2 | 2
Nausea (Gastrointestinal disorders) | 2 | 2
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 2 | 2
Gastric outlet obstruction (Gastrointestinal disorders) | 5 | 2
Radiation gastritis (Gastrointestinal disorders) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 7
Stroke (Nervous system disorders) | 0 | 2
Whipple resection (Surgical and medical procedures) | 2 | 1
Gastrointestinal bleeding (Gastrointestinal disorders) | 5 | 5
Vomiting (Gastrointestinal disorders) | 0 | 1
Perforation (Gastrointestinal disorders) | 0 | 2
Diarrhea (Gastrointestinal disorders) | 5 | 1
Small bowel obstruction (Gastrointestinal disorders) | 2 | 0
Hernia (Gastrointestinal disorders) | 0 | 1
Liver abscess (Hepatobiliary disorders) | 2 | 1
Cholangitis without biliary obstruction (Hepatobiliary disorders) | 1 | 1
Cellulitis (Infections and infestations) | 1 | 0
Fever (Infections and infestations) | 1 | 0
Seizure (Nervous system disorders) | 0 | 1
Change in mental status (Nervous system disorders) | 1 | 0
Spinal surgery for cervical stenosis (Surgical and medical procedures) | 0 | 1
Pulmonary embolus (Vascular disorders) | 1 | 1
Myocardial infarction (Cardiac disorders) | 0 | 1
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Urinary obstruction (Renal and urinary disorders) | 0 | 1
Kidney stone (Renal and urinary disorders) | 1 | 0
Epistaxis (Vascular disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes